CLINICAL TRIAL: NCT01992120
Title: Utility of High-Fidelity Simulation In the Education and Assessment of Residents in the Recognition and Management of the Sepsis Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Key Personnel left institution
Sponsor: NYU Langone Health (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: VA01419
Record Dates: First submitted 2013-10-30; First posted 2013-11-25 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Medical Knowledge; Clinical Performance
Keywords: Simulation; Sepsis; High-fidelity; Severe Sepsis; Septic Shock; Education
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Educational Status; Crisis Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Debriefing of high-fidelity sepsis simulation scenarios (Experimental): First visit:
  * Subjects will fill out a self-assessment focusing on perceptions of their knowledge and ability in the recognition and management of sepsis in hospitalized patient
  * Subjects will be specifically exposed to high-fidelity simulated sepsis scenarios and be debriefed on their performance in these scenarios (intervention)
  * Subjects will take a written test focusing on early recognition and management of sepsis
  * Subjects will receive a didactic teaching session focusing on recognition and management of early sepsis in the hospitalized patient
  In the second visit:
  * Subjects will be exposed to a number of high-fidelity simulated sepsis scenarios and be scored on their performance in management of these scenarios
  * Subjects will take a written test of knowledge focusing on early recognition and management of sepsis
  * Subjects will then be debriefed specifically on their performance in the simulation scenarios
  Interventions: Other: Debriefing of high-fidelity sepsis simulation scenarios
- Debriefing of high-fidelity non-sepsis simulation scenarios (Placebo Comparator): First visit:
  * Subjects will fill out a self-assessment survey of their perceptions of their knowledge and ability in the recognition and management of sepsis in the hospitalized patient
  * Subjects will be exposed to high-fidelity simulation scenarios (non-sepsis) and be debriefed in terms of their performance in these scenarios
  * Subjects will take a written test of knowledge focusing on early recognition and management of sepsis
  * Subjects will receive a didactic teaching session focusing on recognition and management of early sepsis in the hospitalized patient
  In the second visit:
  * Subjects will be exposed to a number of high-fidelity simulated sepsis scenarios and be scored on their performance in management of the scenarios
  * Subjects will take a written test of knowledge focusing on early recognition and management of sepsis
  * Subjects will then be debriefed specifically on their performance in the simulation scenarios
  Interventions: Other: Placebo: Debriefing of high-fidelity non-sepsis simulation scenarios

INTERVENTIONS:
Other: Debriefing of high-fidelity sepsis simulation scenarios — Educational intervention
  Other Names: Education; High-fidelity simulation; Debriefing
  Arms: Debriefing of high-fidelity sepsis simulation scenarios
Other: Placebo: Debriefing of high-fidelity non-sepsis simulation scenarios
  Arms: Debriefing of high-fidelity non-sepsis simulation scenarios

SUMMARY:
The primary objective of the proposed study will be to determine if a multi-modality teaching curriculum utilizing high-fidelity simulation and didactic lecture will result in sustained improvement by internal medicine residents in written knowledge and clinical performance when compared to residents receiving a curriculum utilizing only didactic lecture. The investigators hypothesis is that the addition of high-fidelity simulation to a traditional didactic lecture curriculum will result in sustained and superior written knowledge and practical performance when compared to a group receiving only didactic lecture on the same topic. Specifically, the investigators will be assessing internal medicine resident knowledge and performance in the area of sepsis in the hospitalized patient, and will shape the investigators teaching curriculum around this focus.

DETAILED DESCRIPTION:
This is a randomized prospective single-blinded pilot study. Residents from the internal medicine residency program will be assigned a unique number to de-identify them, and then randomized, stratified by post-graduate year (PGY) level, by random number generator to intervention and control groups. Only de-identified information will be used in subsequent analysis, and no individual results will be used. Residents will not know to which group they have been randomized.

Both the intervention and control groups will take a pre-course survey assessing their level of training, area of specialty/interest, and level of confidence in the recognition and management of sepsis.

Both the intervention and control groups will then be put through 2-4 simulated scenarios using high-fidelity simulation. In the intervention group, these scenarios will be sepsis syndrome scenarios. In the control group, non-sepsis scenarios will be administered.

Immediately following the scenarios, a written knowledge quiz focusing on recognition and management of sepsis will be administered to subjects in both groups.

Following the quiz, there will be a debrief session for subjects in both groups of the simulation scenarios, pointing out what was done correctly and what was not.

There will then be a brief didactic teaching session focusing on recognition and management of sepsis administered to subjects in both groups.

2-4 months later, subjects in both groups will be brought back to the simulation lab and tested on a new identical set of simulated sepsis scenarios. This will be videotaped and scored by an impartial volunteer who will score performance according to a check-list of critical actions. Following the simulated scenarios, the written quiz administered at the first visit will be given again. Subjects in both groups will then get debriefed on their performance.

Data can then be compared between the control and intervention group in terms of written and practical performance. Other potential analyses include before and after performance in the intervention group, comparison between the intervention and control groups, as well as subanalysis by PGY level. Student's paired and unpaired t-test will be the model for statistical analysis, and the investigators will utilize a statistician for data analysis.

In developing and implementing a multi-modality sepsis teaching curriculum, and demonstrating its superiority to a didactic-only curriculum, the investigators hope to justify the permanent implementation of a multi-modality teaching module to educate residents (and other healthcare personnel) which will lead to improved recognition and management of sepsis and improved patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking internal medicine resident trainees

Exclusion Criteria:

* Anyone not meeting inclusion criteria

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Performance on a written assessment of the recognition and management of early sepsis in the hospitalized patient. | 2-4 months after intervention
  Written test
Performance on a practical assessment of the recognition and management of early sepsis in the hospitalized patient. | 2-4 months after intervention
  Graded performance in simulated sepsis scenario utilizing high-fidelity simulation

SECONDARY OUTCOMES:
Self-assessment of knowledge and ability in the recognition and management of early sepsis in the hospitalized patient. | 2-4 months after intervention
  Written self-assessment survey

CONTACTS AND LOCATIONS:
Locations (1):
- VA Harbor Simulation Center, New York, New York, United States